CLINICAL TRIAL: NCT00110695
Title: A Phase 2 Study of Neoadjuvant Chemotherapy With Sequential Weekly Nanoparticle Albumin Bound Paclitaxel (Abraxane) Followed by 5-Fluorouracil, Epirubicin, Cyclophosphamide (FEC) in Locally Advanced Breast Cancer
Brief Title: Therapy With Abraxane and 5-Fluorouracil, Epirubicin, Cyclophosphamide (FEC) for Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-AX-003
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Breast Neoplasms
Keywords: NSABP; Abraxis; Abraxane; Locally advanced breast cancer; Fluorouracil; Epirubicin; Cyclophosphamide; FEC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Nanoparticle albumin bound paclitaxel followed by FEC

INTERVENTIONS:
Drug: Nanoparticle albumin bound paclitaxel followed by FEC — Nanoparticle albumin bound paclitaxel 100 mg/m2 IV for 30 minutes once weekly for 12 weeks followed by FEC (5-FU 500mg/m2 IV push; epirubicin 100 mg/m2 IV over 15 min. [or if given with trastuzumab 75 mg/m2 IV over 15 min.]; cyclophosphamide 500 mg/m2 IV over 30 min.) on Day 1 every 21 days

SUMMARY:
The purpose of this study is to learn how breast cancer tumors respond to a drug called Abraxane followed by a combination of 3 chemotherapy drugs commonly used for breast cancer.

DETAILED DESCRIPTION:
This is a Phase 2, non-randomized study of neoadjuvant treatment with nanoparticle albumin bound paclitaxel (Abraxane) every week for 12 weeks followed by 5-FU, epirubicin, and cyclophosphamide (FEC) every 3 weeks for 4 cycles in women with locally advanced breast cancer. Patients with HER-2 overexpressing breast cancer may receive trastuzumab concurrently with the chemotherapy at the discretion of the investigator. The primary aim of this study is to determine the pathologic complete response rate (pCR) of this sequential regimen.

Patients who achieve clinical complete response (cCR), clinical partial response (cPR), or have resectable stable disease (SD) will undergo surgery. Surgery will consist of modified radical mastectomy or excision of the primary tumor site with clear surgical margins accompanied by axillary staging. Tumor samples taken prior to initiation of treatment will be analyzed for molecular and genetic changes which will be correlated with tumor response.

Patients must have a histologically confirmed diagnosis of breast cancer without documented evidence of distant metastatic disease. Patients with clinical Stage IIB (T3N0 only), IIIA, or IIIB breast cancer will be potential candidates for this trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Diagnosis made by core biopsy or incisional biopsy
* Histologic confirmation of invasive breast cancer
* Clinical staging as IIB (cT3N0 only), IIIA (cT3N1 or cT0-3N2), or IIIB (cT4N0-2)
* ECOG performance 0 or 1
* At the time of entry: *Absolute neutrophil count (ANC) must be greater than or equal to 1200/mm3; *platelet count must be greater than or equal to 100,000/mm3; *hemoglobin must be greater than or equal to 10 g/dl; *serum creatinine must be less than or equal to ULN for the lab.
* The following criteria for evidence of adequate hepatic function must be met: *Total bilirubin must be less than or equal to ULN for the lab unless the patient has a grade 1 bilirubin elevation (> ULN to 1.5 x ULN) due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and *alkaline phosphatase must be < 2.5 x ULN for the lab; and

  *AST must be less than or equal to 1.5 x ULN for the lab.
* MUGA scan or echocardiogram within 3 months prior to entry if: *age greater than or equal to 60, or *history of hypertension, or *plan to receive trastuzumab. For any patient who has a MUGA scan or echocardiogram performed for any reason, the baseline LVEF must be greater than or equal to LLN for the facility performing the procedure and there must be no regional wall abnormalities

Exclusion Criteria:

* Clinical stage IIB disease that is cT2N1.
* Definitive evidence of metastatic disease (M1 by AJCC criteria)
* Prior history of invasive breast cancer in either breast or ductal carcinoma in situ (DCIS) in the ipsilateral breast treated with radiation therapy (patients with a history of lobular carcinoma in situ [LCIS] are eligible).
* Any treatment for the currently diagnosed breast cancer prior to study entry including radiation therapy, chemotherapy, and/or hormonal therapy.
* Pregnancy or lactation at the time of study entry.
* Prior anthracycline or taxane-containing chemotherapy for any malignancy.
* Nonmalignant systemic disease (cardiovascular, renal, hepatic, diabetes, etc.) that would preclude the patient from receiving study treatment or would prevent required follow-up.
* Grade 2 or greater peripheral polyneuropathy at the time of entry.
* Cardiac disease that would preclude the use of anthracyclines or trastuzumab. This includes:

  *myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LV function; *angina pectoris that requires the use of anti-anginal medication; *any history of documented congestive heart failure; *serious cardiac arrhythmia requiring medication; *severe conduction abnormality; *valvular disease with documented cardiac function compromise; or *uncontrolled hypertension defined as blood pressure > 160/100 mm/Hg.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc. (These patients are eligible if this therapy is discontinued prior to randomization.) Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulator (SERM), either for osteoporosis or breast cancer prevention. Patients are eligible only if these medications are discontinued prior to randomization.
* Use of any investigational agent within the month before enrollment in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
pathologic complete response rate in the breast for patients with locally advanced breast cancer (LABC) who receive Abraxane | pCR examined in breast tissue taken at surgery

SECONDARY OUTCOMES:
pathologic complete response rate in the breast and axillary nodes (pCR breast and nodes) in all patients | pCR examined in breast and lymph node tissue taken at surgery
complete clinical response rate (cCR) of the sequential regimen in patients who present with palpable measurable disease | physical exam between the two chemotherapy regimens and at completion of the entire treatment regimen
complete clinical and imaging response rate (ciCR) of the sequential regimen in all patients | physical exam and breast imaging at 3-4 weeks after the last chemotherapy treatment
complete clinical response rate (cCR)of Abraxane in patients who present with palpable measurable disease | physical exam at completion of the Abraxane portion of the treatment regimen
toxicity of the sequential chemotherapy regimen | during treatment and for 3 to 4 weeks after the last chemotherapy cycle
toxicity of the sequential chemotherapy regimen when administered concurrently with trastuzumab | during treatment and for 3 to 4 weeks after the last chemotherapy cycle
2-year progression-free survival | from the first dose of study therapy to first date of disease progression or for a maximum of 24 months from study entry
2-year overall survival (OS) | from the first dose of study therapy to date of death or for a maximum of 24 months from study entry
exploration of molecular and genetic correlates of response | after specimen procurement and continuing after completion of clinical phase of study

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (1):
- NSABP Operations Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Robidoux A, Buyse M, Buzdar A, et al.: Neoadjuvant chemotherapy with sequential weekly nanoparticle albumin-bound paclitaxel (ABI-007, Abraxane®) followed by 5-fluorouracil, epirubicin and cyclophosphamide (FEC) in locally advanced breast cancer (LABC): a phase II trial of the NSABP Foundation research program (FRP). [Abstract] Annual San Antonio Breast Cancer Symposium 3068, 2006.
- [Result] Robidoux A, Buzdar AU, Quinaux E, Jacobs S, Rastogi P, Fourchotte V, Younan RJ, Pajon ER, Shalaby IA, Desai AM, Fehrenbacher L, Geyer CE Jr, Mamounas EP, Wolmark N. A phase II neoadjuvant trial of sequential nanoparticle albumin-bound paclitaxel followed by 5-fluorouracil/epirubicin/cyclophosphamide in locally advanced breast cancer. Clin Breast Cancer. 2010 Feb;10(1):81-6. doi: 10.3816/CBC.2010.n.011. PMID 20133263